CLINICAL TRIAL: NCT05418062
Title: Managing Pain in People With Crohn's Disease: Feasibility Testing of an Acceptance and Commitment Group Therapy Intervention.
Brief Title: Group ACT for CD Pain- a Feasibility Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 314107
Record Dates: First submitted 2022-05-10; First posted 2022-06-14 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-05

CONDITIONS: Chronic Pain; Crohn Disease
MeSH Terms: conditions — Chronic Pain; Crohn Disease | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Masking Description: Not possible die to study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Patients randomised into Group 1 will begin the 8 week group first.
  Interventions: Behavioral: Acceptance and commitment therapy (ACT)
- Control crossover group (Other): Patients randomised into Group 2 will act as the control for the first 8 weeks and then cross over into the intervention arm.
  Interventions: Behavioral: Acceptance and commitment therapy (ACT)

INTERVENTIONS:
Behavioral: Acceptance and commitment therapy (ACT) — 8 weekly 2 hour sessions of ACT group for CD patients with chronic pain. Manual available on request

SUMMARY:
Pain is a common symptom of inflammatory bowel disease (IBD) and has a significant impact on patient quality of life. Pain will frequently be the presenting complaint and is experienced throughout the disease course. Up to 70% of patients experience pain in active disease, and up to half (20-50%) of patients will experience pain in remission.

Pain in IBD is widely recognised as a biopsychosocial construct, with visceral hypersensitivity, as well as depressive symptoms, anxiety, stress and fear avoidance correlating positively with IBD-pain. There is increasing understanding of the psychological interaction and need for psychological management within IBD. Psychological therapies such as Cognitive Behavioural Therapy (CBT) and acceptance and commitment therapy (ACT) have been used widely in other conditions, such as chronic pain, fatigue and irritable bowel syndrome (IBS).

Although neither ACT nor CBT have been used specifically for pain in IBD, ACT has become a regular therapy in the management of chronic pain and a large number of studies have found it to be effective, particularly in relation to improving functioning and decreasing distress, quality of life and physical wellbeing.

This study design is a crossover randomised controlled trial of ACT versus treatment-as-usual (TAU) in people with CD and chronic abdominal pain. The research team aim to assess the feasibility of ACT for reducing the impact of abdominal pain and its associated psychological burden in people with Crohn's disease (CD). The study will investigate the acceptability of ACT to people with CD and chronic pain, specifically testing issues of eligibility, recruitment, retention rates, patient experience and performance of proposed outcome measures. This will inform the design of a subsequent large multi-centre randomised controlled trial (RCT) with long-term follow-up.

DETAILED DESCRIPTION:
Aims:

This study aims to assess the feasibility of ACT for reducing the impact of abdominal pain and its associated psychological burden in people with Crohn's disease (CD). The study will investigate the acceptability of ACT to people with CD and chronic pain, specifically testing issues of eligibility, recruitment, retention rates, patient experience and performance of proposed outcome measures. This will inform the design of a subsequent large multi-centre randomised controlled trial (RCT) with long-term follow-up.

Design and setting:

The design is a crossover randomised controlled trial of ACT versus treatment-as-usual (TAU) in people with CD and chronic abdominal pain. The researchers will invite participants aged 18 and over with a diagnosis of CD attending outpatient clinics at Guy's and St Thomas' NHS Foundation Trust and King's College Hospital NHS Foundation Trust to participate. With ~90 patients with CD attending the clinics each week, this represents one of the largest CD cohorts in the UK. Patients with CD attending the outpatients department will be screened for the presence of chronic pain using standard questionnaires. Individual cases will then be reviewed by a gastroenterologist to assess whether their IBD is stable and they are suitable for the study or whether their pain is part of an acute flare which necessitates a change in medical treatment. Only patients where it is thought pain is part of stable chronic disease will be recruited.

Sample size and recruitment:

This is a feasibility study and power calculations for a treatment effect are not applicable. Based on an expected follow-up rate of at least 75%, a two-sided confidence interval will extend no more than 12.5% of the observed proportion with a sample size of 48 patients, thus providing adequate precision estimates. Based on pilot work in the IBD clinics and our previous experience of running RCTs for psychological therapy in IBD, the researchers conservatively estimate that 25% of people approached will be both willing and eligible to participate. As such, a total of 192 people will be approached to meet the recruitment target. WCD will chair biweekly study meetings where recruitment will be reviewed and intensified if falling behind this trajectory.

Randomisation:

Participants will be randomly allocated (1:1) to the intervention or TAU control group using a web-based randomisation service, which employs block randomisation with randomly varying block sizes. Randomisation will be stratified by male/female sex. The researcher analysing the data will not be able to access the data until final database lock.

Intervention:

Half of the cohort (n=24) will be randomised initially to TAU, which will comprise usual care from the CD team and GP but no specific pain intervention except a CCUK information sheet on pain in CD. After completing 24 weeks of TAU, these patients will then crossover to the intervention.

The other half (n=24) will be randomised initially to the intervention group. In addition to TAU, the intervention group will undergo eight 90-minute sessions of weekly ACT in groups of 8 patients, all led by a single clinical psychologist accredited in ACT. The course is based on contemporary ACT models and tailored toward people with IBD with an emphasis on reducing the impact of pain on functioning and quality of life. The research team will develop a manual and observe the sessions for assessment of fidelity.

The manual will be adapted from one developed by co-applicant AD for use with people with IBD. It will be peer-reviewed by experienced ACT practitioners to ensure adherence to the model. Treatment commences with the therapist aiming to foster the therapeutic alliance; exploring the developing of chronic pain; and explaining the treatment model. Subsequent sessions will include exercises to increase patients' awareness of the long-term consequences of struggling to control pain; their willingness to experience pain; the development of personal value-based goals and their engagement in these. Treatment finishes with a review of progress and plans for barriers in future. Patients will be given weekly homework tasks to develop their individual value-based goals and explore barriers that appear for them. The aim of the sessions is to increase patients' awareness of misplaced control strategies and to relinquish these and to increase their value-based activities.

The therapist will maintain a log of completed and non-completed sessions and any adverse events. The therapist will receive weekly supervision with an experienced ACT therapist (AD) to maintain adherence to the treatment protocol; to discuss issues arising from sessions; and plan for subsequent sessions. Any current treatment for pain will continue and be recorded. Changes to analgesia during the study are not restricted and will likewise be recorded. People randomised initially to the intervention group will not subsequently undergo transfer to the TAU group, as outcomes such as pain may already have been improved by the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of CD according to clinical notes for a minimum of 6 months

Moderate pain, defined as mean score ≥4/10 on both pain severity and pain interference questions the Brief Pain Inventory (BPI) - a validated cut-off to define moderate pain

Duration of pain of at least 3 months

No changes to CD medication made for the previous 2 months

Exclusion Criteria:

* Diagnosis of ulcerative colitis or indeterminate colitis

Known diagnosis of dementia/psychosis or expressing active suicidal ideation on clinical assessment

Currently undergoing other psychological therapy

Primary source of pain is non-abdominal

Non-fluency in verbal English

Pain is identified as a part of acute flare where immediate change in medical treatment is more appropriate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-01-11 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
recruitment rate | Through study completion, an average of 24 weeks
  Do patients want to be recruited/ randomised into the study
retention rate | Through study completion, an average of 24 weeks
  once randomised, do patients continue to engage in the study
completion rate | Through study completion, an average of 24 weeks
  How many patients "complete" the intervention (Attend 5 or more sessions)

SECONDARY OUTCOMES:
Pain severity | Screening, Baseline, Week 8, and 24 after randomisation
  the BPI severity questions assess pain at its "worst," "least," "average," (each over the last 24 hours) and "now" (current pain)
The UK Inflammatory Bowel Disease Quality of Life Questionnaire | Baseline, Week 8, and 24 after randomisation
  Quality of life: the UK IBDQ measures quality of life as measured in several domains: Emotional function, Bowel function, Social Function and Systemic function. Scale: None-> All/ almost all the time. Higher score means Higher level of impact from the condition.
The Inflammatory Bowel Disease-Fatigue questionnaire | Baseline, Week 8, and 24 after randomisation
  This was developed by two of the study investigators (WCD and CN) alongside people with IBD and provides the only validated fatigue scale specific to IBD. Scale 0= None of the time 4= All of the time. Higher score indicates higher levels of Fatigue.
Depression, stress and anxiety: | Baseline, Week 8, and 24 after randomisation
  The Depression Anxiety Stress Scales (DASS-21). Used previously in a study of ACT in IBD, this consists of three 7-item depression, anxiety, and stress survey tools Scale: 0=Did not apply to me at all. 3=Applied to me very much or most of the time. A higher score in each section indicates symptoms.
Pain Acceptance | Baseline, Week 8, and 24 after randomisation
  The Chronic Pain Acceptance Questionnaire (CPAQ-8) which measures acceptance of chronic pain; attempts to avoid or control pain; and the degree of engagement in activities. Scale: 0= Never True, 6= Always True
IBD-Distress | Baseline, Week 8, and 24 after randomisation
  The IBD-Distress Scale (IBD-DS), this 28-item scale (co-developed by WCD and CN) has good face and content validity and excellent internal consistency. Yes/ No , If Yes, Scale: 1= mildly distressing, 6=Highly Distressing. Higher scores indicates higher levels of distress.
Treatment evaluation | Post treatment Week 8, or 24
  numerical ratings reflecting how interesting, successful and logical participants perceived the treatment to be on a scale of 0-10.
Impairment in functioning:. | Baseline, Week 8, and 24 after randomisation
  The Work and Social Adjustment Scale (WSAS), which provides a 5-question index of impairment in functioning attributable to an identified problem. Scale 0= Not at all, 8=Very severely.
Pain Interference | Screening, Baseline, Week 8, and 24 after randomisation
  the mean score on the pain interference questions on the BPI. This measures the degree to which pain has interfered with 7 daily activities (general activity, walking, work, mood, enjoyment of life, relations with others and sleep). This mean score will be used if more than 50% of the total items have been completed on a given administration. Scale: 0= Does not interfere, 10=Completely interferes
SIMPLE INDEX OF CROHN'S DISEASE ACTIVITY (Harvey & Bradshaw 1980) | Screening, Baseline, Week 8, and 24 after randomisation
  A) General Wellbeing: (Very well/slightly below par/poor/very poor/ Terrible), B) Abdominal pain (None, Mild, moderate, severe), C) Number of liquid stools per day:..... D) Abdomen feels Lumpy ( None, Dubious, Definite, Definite and tender), E) Complications please tick all that apply: Painful joints/ arthritis, Anal fissure/ fistula/ abcess, Mouth ulcers, Skin nodules or ulcers, Eye pain or inflammation (Red eyes), Liver Problems (e.g primary sclerosing cholangitis)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Wladyslawa Czuber-Dochan, Principal Investigator — KCL
Locations (1):
- Natalie Watson, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391